CLINICAL TRIAL: NCT01351701
Title: An Observational, Prospective, Multicentre Study in Eastern India to Understand the Bacteriological Epidemiology in Diabetic Foot and Sensitivity Pattern of Antibiotics Along With the Pattern of Empirical Therapy
Brief Title: Bacteriological Study of Diabetic Foot and Antibiotic Sensitivity Pattern in Eastern India
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Valley Hospital, Guwahati (Other)
Responsible Party: DR SUDHIR KR JAIN drsudhirguw@gmail.com 09864062104, Dr Sudhir jain, Sun valley Hospital, Guwahati
Other Study IDs: Sunvalley Diabetic Foot Study
Record Dates: First submitted 2011-04-29; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-04

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot; Bacteriological epidemiology; Wagner's Grading; eastern India
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The pattern of organism causing diabetic foot infection are presumed to vary from location to location depending on the antibiotic prescription practice, geographical locations, environmental variations and therapeutic interventions for various patients. Our hypothesis is look to finding out common similarities with diversified subgroups spread across various geographical locations of eastern part of India, thus to create a data base for treating patient with diabetic foot infections.The sensitivity pattern is anticipated to be different from institution to institutions and place to place but the gross sensitivity data of local pathogen could guide physician for choosing right empirical antibiotic. Practice guideline could be postulated from the collated data of distribution of pathogens, their sensitivity pattern as well as co-morbid conditions of the sufferers.

ELIGIBILITY:
Inclusion Criteria:

* diabetic foot patients with Wagner's grade 2 or more foot infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Mixed-Rural/Urban in three eastern states of India
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Epidemiological pattern of diabetic foot infection in eastern India | One year
Sensitivity of isolated organisms to antibiotics | one year
Risk factors associated with different grades of severity of DFI | one year

SECONDARY OUTCOMES:
To record prevailing management practices of diabetic foot infection in terms of disease, antibiotic practice, practice of supportive and surgical care. | one year
Common empiric antibiotic therapies used in management of DFI | one year
Percentage sensitivity to different empiric antibiotics | one year

CONTACTS AND LOCATIONS:
Overall Officials: DR SUDHIR Kr JAIN, MS (Surgery), Principal Investigator — Sun Valley Diabetic Care and Research Centre
Locations (1):
- Sun Valley Diabetic Care And Research Centre, Guwahati, Assam, India